CLINICAL TRIAL: NCT01906944
Title: Ultrasound Guided Transversus Abdominis Plane Block vs. Trigger Point Injection for Abdominal Wall Pain: A Randomized Comparative Trial
Brief Title: Ultrasound Guided Transversus Abdominis Plane (TAP) vs. Trigger Point Injection (TPI) for Abdominal Wall Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Susan M. Moeschler, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-004223
Record Dates: First submitted 2013-07-01; First posted 2013-07-24 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Pain
Keywords: trigger point injection; transversus abdominis plane; abdominal wall pain
MeSH Terms: conditions — Abdominal Pain | interventions — Bupivacaine; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trigger point injection (Active Comparator): Trigger point injection under ultrasound guidance into the fascial layer above the external oblique or rectus muscle, whichever corresponds to patient's identifiable trigger point. The injectate will include 5 ml of bupivacaine 0.25% mixed with triamcinolone 20 mg.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Triamcinolone
- Transversus abdominis plane block (Active Comparator): Injection into transversus abdominis plane layer under ultrasound guidance on the affected side along the mid-axillary line. The injectate will include 10 ml of bupivacaine 0.25% mixed with triamcinolone 20 mg.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Triamcinolone

INTERVENTIONS:
Drug: Bupivacaine 0.25% — Bupivacaine is a local anaesthetic drug belonging to the amino amide group.
  Other Names: Marcain; Marcaine; Sensorcaine; Vivacaine
Drug: Triamcinolone — Triamcinolone is a long-acting synthetic corticosteroid.
  Other Names: KENALOG-40

SUMMARY:
Patients with chronic abdominal pain- with a component of abdominal wall pain- are often treated with trigger point injections. This study will help to determine if a block within the transversus abdominis plane (TAP) will provide superior analgesic benefit to a trigger point injection as therapy for these patients.

DETAILED DESCRIPTION:
Only patients referred to the Pain Clinic for abdominal trigger point injections for abdominal wall pain will be considered for study recruitment.

Following informed consent, patients will complete a baseline questionnaire in the Pain Clinic which gathers basic demographic data, pain scores and functional scores. Patients will be randomized to receive either a TAP injection or a TPI. Because the TAP injection involves a larger area to be anesthetized, a larger volume of medication will be used.

Thirty minutes after the injection, a sensory exam will be performed on the patient to determine the level of block. At one week, one month, three months and six months after the injection, a staff member will telephone the patient to assess how they are doing. The call will take approximately 10 minutes and will consist of relaying a pain score as well as daily functioning and sleep questions.

Subjects are responsible for all clinical costs associated with the injection.

There is no remuneration offered for study participation.

ELIGIBILITY:
Inclusion Criteria:

Only patients referred to Pain Clinic for a trigger point injection.

* Non-cancer pain greater than 3 months duration.
* Unilateral abdominal pain.
* Positive Carnett's sign (A test in which acute abdominal pain remains unchanged or increases when the muscles of the abdominal wall are tensed.)
* An identifiable abdominal trigger point.

Exclusion Criteria:

* History of chronic psychotic disorder.
* History of dementing illness.
* Active abdominal visceral disease as a known contributor of the pain.
* Abdominal surgery in the past 6 months.
* More than one trigger point.
* Abdominal wall hernias.
* BMI>40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Change in Mean Numerical Pain Score | baseline to 6 months
  Pain intensity will be assessed using the 11-point Numerical Pain Score questionnaire where "0" denotes no pain and "10" signifies the most intense pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Moeschler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Moeschler SM, Pollard EM, Pingree MJ, Pittelkow TP, Bendel MA, Mauck WD, Watson JC, Eldrige JS, Loftus CG, Hooten WM. Ultrasound-guided transversus abdominis plane block vs trigger point injections for chronic abdominal wall pain: a randomized clinical trial. Pain. 2021 Jun 1;162(6):1800-1805. doi: 10.1097/j.pain.0000000000002181. PMID 33433147
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials